CLINICAL TRIAL: NCT06875115
Title: Evaluation of the Efficacy of Laser Acupuncture on Uremic Pruritus-Randomized Controlled Trial Double Blind
Brief Title: Evaluation of the Efficacy of Laser Acupuncture on Uremic Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B11301036
Record Dates: First submitted 2024-08-23; First posted 2025-03-13 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Uremia
Keywords: uremia
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser acupuncture on acupoint (Active Comparator): The experimental group is a powered, functional laser device,
  Interventions: Device: laser acupuncture
- shame laser on acupoints (Placebo Comparator): the control group is a non-functional laser device that does not emit light and has no therapeutic effect.
  Interventions: Device: laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — laser acupuncture on acupoints

SUMMARY:
Sixty patients were randomly assigned to either the experimental group (n=30) receiving laser acupuncture or the control group (n=30) receiving sham laser acupuncture. Treatment sessions were conducted during dialysis sessions. The experimental group received laser acupuncture at Xuehai, Quchi, and Bai Chongwo acupoints three times per week for four weeks. The control group received sham laser acupuncture at the same acupoints. The 5-D Pruritus Scale and DLQI were used to assess pruritus severity before and after the intervention.

DETAILED DESCRIPTION:
The subjects were divided into two groups to investigate whether laser acupuncture can improve uremic pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years.
* Intact parathyroid hormone (iPTH) levels < 68 pg/mL (patients with -thyroidectomy excluded).
* Urea nitrogen (BUN) clearance rate (Kt/V) ≥ 1.2 at each dialysis session.
* Serum phosphate levels < 5.5 mg/dL.
* Receiving hemodialysis three times weekly for at least three consecutive months.
* No history of acute illnesses like infections or cardiovascular disease.
* Avoiding a high-phosphorus diet.
* Adjusting dialysate calcium concentration to 8.6-10 mg/dL.
* Replacing the artificial kidney or increasing dialysis blood flow

Exclusion Criteria:

* Pregnant or nursing.
* History of photosensitivity.
* Recent use of systemic or local medications for pruritus (e.g., immunosuppressants, opioid agonists/antagonists, glucocorticoids, antihistamines, ultraviolet B therapy).
* Hepatobiliary dysfunction based on medical history and liver function tests.
* Malignancies.
* Other itchy skin conditions diagnosed by a dermatologist.
* Wounds near acupuncture points, contraindicating laser acupuncture

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2025-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying-HSU Juan, doctor, Study Chair — doctor
Locations (1):
- Dalin Tzu Chi Hospital, Dalin, Chiayi, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the hemodialysis center of Dalin Tzu Chi Hospital between January 2024 and December 2024. Eligible patients were screened based on inclusion/exclusion criteria during routine dialysis visits. Written informed consent was obtained prior to enrollment. A total of 60 participants met eligibility criteria and agreed to join the study.
Pre-assignment Details: All 60 consented participants completed baseline assessment and proceeded to randomization without exclusions. No participants withdrew or were removed prior to group assignment.
Groups:
- Sham Laser: Participants received sham laser acupuncture at the same acupoints (Quchi, Xuehai, Baichongwo) using identical device appearance and procedure, without active laser output. Frequency and duration matched the active group.
- Laser Acupuncture: Participants received low-level laser acupuncture delivered to Quchi (LI11), Xuehai (SP10), and Baichongwo (EX-LE4) bilaterally, three times per week for 4 weeks during routine hemodialysis sessions. Laser parameters were standardized for all treatments.
Period: Overall Study
Arm/Group | Sham Laser | Laser Acupuncture
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Laser | Laser Acupuncture | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.27 (12.39) | 59.20 (11.52) | 58.24 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Title: Evaluation of the Efficacy of Laser Acupuncture on Ureimc Pruritus
Description: The severity of uremic pruritus was assessed using the 5-D Itch Scale, a validated instrument that measures itch duration, degree, direction, disability, and distribution. The total score ranges from 5 to 25, with higher scores indicating worse pruritus. Measurements were taken at baseline and at week 4 after completion of the laser acupuncture or sham intervention.
Time Frame: A 4-week timeframe from enrollment to treatment completion.
Measure: Mean (Standard Deviation); unit: points
Groups:
- Laser Acupuncture: Participants received laser acupuncture at Quchi (LI11), Xuehai (SP10), and Baichongwo (EX-LE4) twice weekly for 4 weeks.
- Sham Laser: Participants received sham laser acupuncture at the same acupoints with an inactive laser device twice weekly for 4 weeks.
Arm/Group | Laser Acupuncture | Sham Laser
Number analyzed (Participants) | 30 | 30
points
  baesline | 18.13 (3.71) | 17.47 (3.58)
  Week 4 | 10.20 (4.96) | 17.10 (3.72)
Statistical Analysis 1: Comparison: Laser Acupuncture vs Sham Laser; Primary Outcome Analysis; Test type: Superiority — The primary outcome (5-D Itch Scale score) will be analyzed by comparing the change from baseline to 4 weeks between the laser acupuncture group and the sham laser group. Continuous variables will be summarized as mean ± standard deviation. Between-group comparisons will be performed using independent t-tests or Mann-Whitney U tests, as appropriate. A two-sided p value < 0.05 will be considered statistically significant; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: From baseline to week 4 during the intervention period.
Groups:
- Sham Laser: Participants received sham laser acupuncture at Quchi (LI11), Xuehai (SP10), and Baichongwo (EX-LE4) using a device with no laser output.
- Laser Acupuncture: Participants received active laser acupuncture at Quchi (LI11), Xuehai (SP10), and Baichongwo (EX-LE4) using a low-level laser device delivering therapeutic output during each session.
Arm/Group | Sham Laser | Laser Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
This study was conducted in a single center with a relatively small sample size, which may limit the generalizability of the findings. The follow-up period was short (4 weeks), and longer-term effects of laser acupuncture on uremic pruritus could not be evaluated. The study population consisted of stable hemodialysis patients, and results may not apply to other patient groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT06875115/Prot_SAP_000.pdf